CLINICAL TRIAL: NCT01250704
Title: Inherited Myokymia: A Clinical and Genetic Study of a Family
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Department of Medical Research, China Medical University Hospital
Other Study IDs: DMR99-IRB-190
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2010-11

CONDITIONS: A Study of Clinical and Genetic Mutations in a Family of Neuromyotonia, so Called Isaac's Syndrome
Keywords: Neuromyotonia, Isaac's syndrome; Peripheral nerve hyperexcitability; Myokymia; Potassium channelopathy
MeSH Terms: conditions — Isaacs Syndrome; Myokymia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Genomic DNA was extracted from each patient's peripheral blood leukocytes using Genomaker DNA extraction kit (Blossom, Taipei, Taiwan). The complete KCNA1 coding region, including the intron/exon boundaries, was amplified according to the procedure reported by Imbrici et al
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Neuromyotonia (NMT), so called Isaac's syndrome, is a rare disorder in which hyperexcitability of peripheral motor nerves leads to intermittent muscle contractions. It is characterized by muscle twitching at rest (visible myokymia), cramps, hyperhidrosis, paraesthesiae, mild muscle weakness. and impaired muscle relaxation, or pseudomyotonia. Electromyographic recording is a key diagnostic tool in detecting myokymia and neuromyotonia. Pathophysiology of neuromyotonia is claimed to be related immune disorder, autoimmune anti-voltage-gated potassium-channel antibodies and genetic mutation in potassium channel. KCNA1 (Kv1.1) mutation was mostly reported in a autosomal dominant trait. In the present study, we report a family affected with myokymia，worsening with elevated body temperature, febrile illness or spicy food. How the change in temperature influence clinical features of channelopathies is an interesting topic. Variant clinical severity of family members are recorded. The index patient has possible autoimmune mechanism involvement because of his clinical feature of myasthenia gravis with thymoma and hyperthyroidism. Further analyzing the genetic mutation in potassium channelopathy may provide researchers some pathophysiological insight into the Isaac's syndrome.

ELIGIBILITY:
Inclusion Criteria:

* The disease was initially diagnosed of Isaacs syndrome by two neurologist(Dr Tsai and Dr Yang). We will recruit family members of diseased patient and normal subjects for clinical, electromyographic and genetic studies.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We interview and examine the family members directly at our hospital and home visit or indirectly by telephone visit.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ting Hsu, MD, Study Director — China Medical University Hospital
Locations (3):
- Taiwan (3):
  - China medical university hospital, Taichung, Taiwan
  - China Medical University Hospital, Taichung
  - China medical university hospital, Taichung